CLINICAL TRIAL: NCT07301918
Title: Evaluation of the Effects of the Leaf Expander Versus Hyrax Expander in Mixed Dentition Patients With Posterior Crossbite: A Randomized Clinical Trial.
Brief Title: Leaf Expander Versus Hyrax Expander in Mixed Dentition Patients With Posterior Crossbite.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura Mohamed Hamza Hassan Saleh, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24619942
Record Dates: First submitted 2025-11-21; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Posterior Crossbite; Maxilla; Hypoplasia
Keywords: expander; maxillary transverse deficiency; posterior crossbite; mixed dentition
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Banded Leaf expander supported on the maxillary first permanent molars (Experimental): 9mm leaf expander delievering 900 gm force will be supported on the upper first permanent molars with the appliance arm extending to the canines
  Interventions: Device: The Leaf expander
- Banded Hyrax expander supported on the maxillary first permanent molars (Active Comparator): 9mm Hyrax expander will be supported on the upper first permanent molars with the appliance arm extending to the canines
  Interventions: Device: Hyrax expander

INTERVENTIONS:
Device: The Leaf expander — The Leaf expander incorporates Nickel Titanium springs that will not require the patients' home activation
  Arms: Banded Leaf expander supported on the maxillary first permanent molars
Device: Hyrax expander — Hyrax expander incorporates a screw that requires the patients' home activation
  Arms: Banded Hyrax expander supported on the maxillary first permanent molars

SUMMARY:
Design: Two-arm parallel randomized clinical trial in mixed dentition (6-12 years).

Arms: (1) 9 mm, 900 g leaf expander; (2) 9 mm Hyrax expander. Follow-up: From appliance insertion → completion of intended expansion → 6-month retention.

Primary outcome: Pain perception during the first 7 days post-insertion (daily patient-reported scale).

Secondary outcomes: Skeletal and dental changes on CBCT.

DETAILED DESCRIPTION:
Participants receive a banded maxillary expansion appliance cemented to maxillary first permanent molars, assigned to:

Leaf expander arm: Nickel-titanium leaf-spring expander, 9 mm screw, delivering force of ~900 g.

Hyrax expander arm: Conventional tooth-borne jackscrew expander, 9 mm screw. Standard activation: two turns per week.

Retention: Both appliances kept passively in situ for 6 months of retention following achievement of planned expansion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Mixed dentition stage
* Unilateral or bilateral posterior crossbite.
* Patients in prepubertal stage with cervical vertebral maturation stage 1-3.
* Fully erupted maxillary and mandibular permanent first molars.
* Skeletal class I or II.

Exclusion Criteria:

* Previous orthodontic treatment.
* Missing teeth.
* Inadequate oral hygiene.
* Patients with bad oral habits.
* Patients with medical conditions.
* Patients with cleft lip and palate.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain perception | first week after appliance insertion
  Pain perception during the first week after insertion using Wong-Becker faces scale with minimum value of zero and maximum value of ten, ten score represents the worst pain percieved.

SECONDARY OUTCOMES:
skeletal expansion | 6 months post expansion
  skeletal expansion using Cone Beam Computed Tomography skeletal expansion: linear distances of the midpalatal suture opening measured in mm between the pre- and post-axial cuts of the CBCT
dental tipping | 6 months post-expansion
  Angular measurement of upper first molars angulation measured in degrees between pre- and post-coronal cuts of the CBCT